CLINICAL TRIAL: NCT00637416
Title: The Effect of Dietary Control Alone Versus Dietary Control Plus Use of Proton Pump Inhibitors to Treat Pediatric Hoarseness
Brief Title: Dietary Control Alone Versus Dietary Control Plus Use of Proton Pump Inhibitors to Treat Pediatric Hoarseness
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: University of Kansas Medical Center (Other)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10720
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Dysphonia
Keywords: horseness
MeSH Terms: conditions — Dysphonia | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole and dietary control (Active Comparator): Lansoprazole and dietary control
  Interventions: Drug: Lansoprazole
- Placebo and dietary control (Placebo Comparator): Dietary control and placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 30 mg taken by mouth daily for 3 months
  Other Names: Prevacid
  Arms: Lansoprazole and dietary control
Other: Placebo — placebo taken by mouth daily for 3 months
  Arms: Placebo and dietary control

SUMMARY:
This study will examine whether lansoprazole (Prevacid) and dietary control versus dietary control alone will improve pediatric hoarseness symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children with a diagnosis of dysphonia age 3-18 years.
2. Dysphonia must be present for at least one month duration.
3. May have vocal cord nodules present.
4. Pre-enrollment flexible fiberoptic laryngoscopy must not show any potentially life-threatening cause, including but not limited to laryngeal papillomatosis, congenital glottic webs, vocal cord paralysis, or benign and malignant neoplasms.
5. Must be able to cooperate with recording of voice for analysis(3 seconds of sustained vowel).
6. Caregiver must be able to read, write, and understand English.
7. Patient with history of diagnosed asthma must have their asthma well controlled and treated at the time of enrollment for study.

Exclusion Criteria:

1. Dysphonia must not be due to a potentially life-threatening cause, such as laryngeal papillomatosis, congenital glottic webs, vocal cord paralysis, or benign and malignant neoplasms. This will be determined by visualization with flexible fiberoptic laryngoscopy.
2. Dysphonia must not be due to an acute upper respiratory infection.
3. Must not have been treated with proton pump inhibitor medication in the past 12 months.
4. Inability of child to cooperate with recording of voice for analysis.
5. Inability of caregiver to read, write, and understand English.
6. Mental retardation, cognitive impairment, or developmental delay.
7. History of allergic reaction of any kind to lansoprazole or any other proton pump inhibitor.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Wei, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lansoprazole and Dietary Control | Placebo and Dietary Control
Started | 4 | 5
Completed | 3 | 3
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Unable to take study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lansoprazole and Dietary Control | Placebo and Dietary Control | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Condition Over Treatment Period
Description: Change measured using voice assessment protocol-Grade, Roughness, Breathiness, Asthenia, Strain (GRBAS).
Time Frame: 3 months
Population: Study was stopped early, data were not collected, and zero participants were analyzed.
Arm/Group | Lansoprazole and Dietary Control | Placebo and Dietary Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Lansoprazole and Dietary Control | Placebo and Dietary Control
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes